CLINICAL TRIAL: NCT03556605
Title: Tu Salud Randomized Controlled Partial Cross-over Study in Patients With Diabetes in an Underserved Population
Brief Title: Tu Salud (Your Health) Randomized Control Study in Patients With Diabetes Using a Mobile App.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LifeScan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PR3170365
Record Dates: First submitted 2018-05-29; First posted 2018-06-14 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Other): A target of 100 subjects will be enrolled in the Intervention arm using the OneTouch Reveal® Mobile APP system
  Interventions: Other: OneTouch Reveal® Mobile APP system
- Control Arm. (Other): A target of 50 subjects will be enrolled in the Control intervention arm. Subjects continue to use their current Blood Glucose Monitor without connection to mobile diabetes apps.
  Interventions: Other: Current Blood Glucose Monitor

INTERVENTIONS:
Other: OneTouch Reveal® Mobile APP system — Improved glycemic control in people with diabetes using the OneTouch Verio® Flex Blood Glucose Monitor and the OneTouch Reveal® Mobile APP system (intervention group) compared to subjects continuing to use their own Blood Glucose Monitor without connection to mobile diabetes apps (control group).
  Arms: Intervention Arm
Other: Current Blood Glucose Monitor — Subjects continue to use current Blood Glucose Monitor without connection to mobile diabetes apps.
  Arms: Control Arm.

SUMMARY:
The study seeks to demonstrate the clinical value and user acceptance of the Bluetooth enabled OneTouch Verio® Flex meter (Flex) used in combination with the OneTouch Reveal® Mobile APP to support overall diabetes care, glycemic control and patient reported outcomes in patients with diabetes in an undeserved population.

DETAILED DESCRIPTION:
This is a parallel arm, open-label, randomized controlled, partial cross-over study. Subjects will be randomized into intervention group or control group in a 2:1 ratio. Intervention group will use the Flex blood glucose meter and OneTouch Reveal Mobile App and receive text messages every 2 weeks from the Health Care Professional for 12 weeks. The intervention group will continue under the same conditions until 24 weeks to explore durability of effects. The control group will use their own blood glucose meter without connectivity to a diabetes app for the first 12 weeks of the study. At that point, control group subjects will cross-over to the same treatment as the intervention group for an additional 12 weeks.

A target of 100 subjects will be enrolled in the Intervention arm and a target of 50 subjects will be enrolled in the Control arm. Randomization will be stratified based on type of diabetes (Type 1 or Type 2) and A1c (above or below 9.0%). Each subject will attend visits at Screening/Baseline, 12 weeks and 24 weeks after Baseline. In most cases, Screening and Baseline will occur on the same day.

Study Periods

The study will be conducted in the following periods:

Visit 1 (Screening/Baseline): All screening procedures will be performed including informed consent, demographics, medical history, a capillary blood draw for POC A1c determination and evaluation of entrance criteria. If subject A1c meets inclusion criteria and subject meets all other inclusion criteria and none of the exclusion criteria, subject will be randomized into one of two arms via randomization scheme. The time of randomization becomes Day 1.

Visit 2 (Week 12 ± 7 days): A capillary blood draw will be performed for measurement of POC A1c. The HCP will discuss diabetes management progress with all subjects: for the control group based on their own meter data; for the intervention group, the HCP will download SMBG data from Flex meters and discuss diabetes management based on OTRM APP and Flex meter information. The HCP will review and consider if the glucose range limits on the Flex meter and/or OTRM need to be updated. Intervention subjects will continue in the same group for an additional 12 weeks. Control subjects will be switched to Flex and OTRM for 12 weeks.

Visit 3 (Week 24 ± 7 days): A capillary blood draw will be performed for measurement of POC A1c. The HCP will download SMBG data from all Flex meters. Subjects will return study materials.

ELIGIBILITY:
Inclusion Criteria:

* Male or female , at least 18 years old.
* Has an A1c ≥7.5 at screening visit
* It is medically appropriate in the opinion of the investigator for the Subject to attempt to achieve a level of glycemic control in line with the ADA guidelines on glycemic recommendations (<7.0% A1c, pre-prandial capillary glucose of 70-130 mg/dl and peak post-prandial glucose of <180 mg/dl)
* Diagnosed with T2D or T1D for ≥ 3 month before screening
* Currently performing SMBG at home for diabetes management decisions and willing to perform SMBG ≥ 1 per day if subject has T2D and is on oral antihyperglycemic (AHA) agents and/or non-insulin injectable (e.g. GLP-1) only; test ≥ 2 times per day if on basal insulin or premixed insulin; and test ≥ 3 times per day if subject has T2D and is on multiple daily injections (MDI) or subject has T1D
* Willing to receive (and send, if necessary) text messages every 2 weeks throughout the study using a smartphone. (note: this inclusion criteria applies to all subjects regardless of whether they are subsequently randomized to control or intervention arms)
* Is in an area that can send and receive text messages and has access to a phone signal to use the network as required
* Willingness to notify the study staff if they become pregnant during the study
* Able to communicate in English or Spanish, and able to understand and sign the required study documents;
* Sign an informed consent document indicating they understand the purpose and procedures of the study

Exclusion Criteria:

* Unlikely to be compliant with the currently prescribed diabetes regimen, in the opinion of the study staff
* Subject is pregnant
* Currently using OneTouch Verio® Flex at home for routine glucose testing
* Currently using OneTouch Reveal app
* Currently using a continuous glucose monitor (CGM) or insulin pump
* Has unstable (rapidly progressing) retinopathy that in the opinion of the study staff may require surgical treatment (including laser photocoagulation) during the study
* Is currently on or received treatment during the past 3 months with the following medications: Systemic corticosteroids or anti-psychotic drugs
* Is currently psychiatrically unstable in the opinion of the study staff
* Has known clinically significant and/or unstable medical conditions which, in the opinion of the study staff, could interfere with participation in the study, including:
* Cardiovascular disease
* Hematological disease
* Hepatic disease.
* Gastrointestinal disease
* Endocrine/metabolic disorders
* Neurologic disease
* History of major surgery within 3 months
* Has had any condition that in the opinion of the study staff that would complicate or compromise the study, or the wellbeing of the Subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-09-15 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in A1c from baseline at 12 weeks in intervention group compared to control group. At this point, control group subjects will cross-over to the same treatment as the intervention group for an additional 12 weeks. | Each subject will attend visits at Screening/Baseline, 12 weeks and 24 weeks after Baseline.
  The primary objective is to demonstrate improved glycemic control in people with diabetes using the OneTouch Verio® Flex Blood Glucose Monitors and the OneTouch Reveal® Mobile APP system (intervention group) compared to subjects continuing to use their own Blood Glucose Monitor without connection to mobile diabetes apps (control group).

CONTACTS AND LOCATIONS:
Overall Officials: Frederico Ceppa, Principal Investigator — La Comunidad Hispana Health Center
Locations (1):
- La Comunidad Hispana (LCH) Health Center, West Chester, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No